CLINICAL TRIAL: NCT00195442
Title: Pharmacovigilance Evaluation Of Refacto In Usual Care Settings
Brief Title: Study Evaluating Refacto For Pharmacovigilance
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Other Study IDs: 3082A-100690
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2011-02-07 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with Hemophilia A
  Interventions: Drug: Moroctocog alfa

INTERVENTIONS:
Drug: Moroctocog alfa — Patients will be treated in accordance with the requirements of the labeling of ReFacto (Moroctocog alfa) in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: ReFacto

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of treatment with ReFacto under conditions of routine therapy. Furthermore a continuous benefit/risk assessment will be done.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of Hemophilia A

Exclusion Criteria:

* Contraindications according to Summary of Product Characteristics

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 1999-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Pfizer Investigational Site, Vienna, Vienna, Austria
- Germany (24):
  - Pfizer Investigational Site, Berlin, Germany
  - Pfizer Investigational Site, Wiesbaden, Germany
  - Pfizer Investigational Site, Frankfurt am Main, Hesse
  - Pfizer Investigational Site, Giessen, Hesse
  - Pfizer Investigational Site, Hanover, Lower Saxony
  - Pfizer Investigational Site, Rostock, Mecklenburg-Vorpommern
  - Pfizer Investigational Site, Bonn, North Rhine-Westphalia
  - Pfizer Investigational Site, Halle, Saxony-Anhalt
  - Pfizer Investigational Site, Stadtroda, Thuringia
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bermen
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Frankfurt A. M.
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Homburg
  - Pfizer Investigational Site, Klipphausen
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Potsdam
  - Pfizer Investigational Site, Schwerin
  - Pfizer Investigational Site, Ulm

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082A-100690&StudyName=Study%20Evaluating%20Refacto%20For%20Pharmacovigilance

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 288 participants were observed during the study in 48 centers (44 Germany and 4 Austria) from time of First subject first visit May 1999 to Last subject last visit January 2010.
Pre-assignment Details: The study was terminated January 2010 due to the introduction of a successor product ReFacto® AF.
Groups:
- ReFacto (Moroctocog Alfa): B-domain deleted, recombinant factor VIII (BDDrFVIII) for participants with Hemophilia A in usual health care settings.
Period: Overall Study
Arm/Group | ReFacto (Moroctocog Alfa)
Started | 288
Completed | 152
Not Completed | 136
Not completed — Less than expected therapeutic effect | 38
Not completed — Lost to Follow-up | 27
Not completed — Switch to other Factor VIII preparation | 23
Not completed — Intermittent product shortage | 21
Not completed — Death | 7
Not completed — No reason specified | 4
Not completed — Poor cooperation | 2
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 288
Age, Customized [Number; unit: participants]
  Children < 18 years of age | 106
  Adults ≥ 18 years of age | 182
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 288

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Bleeding Episodes Per Patient Year
Description: Participants with hemophilia A suffer from a hereditary lack of blood clotting factor VIII. As a consequence, the ability of the blood to coagulate is reduced and bleedings at any site or organ of the body may occur after minor injury or even spontaneously. Predominantly, joints, muscles, and internal organs are affected by bleeding complications. Participants reported the occurrence of each bleeding episode while on study. The bleeding rate for each participant was calculated by number of reported episodes per years on study.
Time Frame: Baseline up to a mean duration of 54 months
Population: Total population for efficacy analysis included all participants with submitted diary cards and severe haemophilia.
Measure: Mean (Standard Deviation); unit: episodes per year
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 192
episodes per year | 13.41 (14.67)

2. Primary Outcome: Mean Number of Bleeding-related Exposure Days Per Patient Year
Description: Exposure days are the number of days of treatment with ReFacto.
Time Frame: Baseline up to a mean duration of 54 months
Population: Total population for efficacy analysis included all participants with submitted diary cards and severe haemophilia.
Measure: Mean (Standard Deviation); unit: days per year
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 192
days per year | 20.58 (21.39)

3. Primary Outcome: Mean Number of Exposure Days Per Patient Year
Description: Exposure days are the number of days of treatment with ReFacto.
Time Frame: Baseline up to a mean duration of 54 months
Population: Total population for efficacy analysis included all participants with submitted diary cards and severe haemophilia.
Measure: Mean (Standard Deviation); unit: days per year
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 192
days per year | 126.76 (68.81)

4. Secondary Outcome: Number of Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs are any undesired side effect which occurred in a participant undergoing study treatment independent of whether a correlation with study treatment was suspected or not. SAEs are undesired events which were lethal or life-threatening, made hospitalization or extension of hospital stay necessary, lead to permanent damage with handicap (inability to work), as well as congenital anomalies, malignant disease, or overdosing. Also presence of inhibitors, thrombotic events, erythrocyte agglutination, allergic reactions, less than therapeutic effect, and inhibitor development were considered SAEs.
Time Frame: Baseline up to a mean duration of 54 months
Population: Safety population includes all subjects with a baseline visit; (n)=number of participants with events.
Measure: Number; unit: events
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 288
events
  Non-serious Adverse Events (n=118) | 668
  Serious Adverse Events (n=141) | 291

5. Secondary Outcome: Number of Participants With de Novo Inhibitor Formation
Description: The applied criteria of clinical relevance for de novo inhibitor formation was defined as normal Factor VIII dosage was ineffective to control a bleeding, control of bleeding episodes required increasing Factor VIII dosage, change of concentrate type (administration of activated Prothrombin-Complex Concentrate [aPCC] or recombinant Factor VII [rFVII ]) was needed to stop a bleeding, or change of therapy strategy (intensive prophylaxis or Immune Tolerance Induction [ITI]) was required.
Time Frame: Baseline up to a mean duration of 54 months
Population: Safety population includes all subjects with a baseline visit.
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 288
participants | 7

6. Secondary Outcome: Mean Annual ReFacto Consumption Per Patient Year
Description: ReFacto administered as International Units (IU) according to the physician's decision following the drug's summary of product characteristics (SPC) and according to usual care principles.
Time Frame: Baseline up to a mean duration of 54 months
Population: Total population for efficacy analysis included all participants with submitted diary cards and severe haemophilia.
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 192
International units per year | 204509 (221723)

7. Secondary Outcome: Number of Participants for Physicians' Assessment of Satisfaction With Treatment Success
Description: Subjective assessment by the physician to evaluate treatment success (i.e., control of bleeding, Factor VIII consumption, treatment efficacy and tolerance, handling of preparation, and days missing from work or school). Physician rated assessment could be categorized as Very satisfied, Satisfied, Unsatisfied, or Very unsatisfied; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: Safety population includes all subjects with a baseline visit. N=participants with evaluable data; last measurement available.
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 169
participants
  Very satisfied | 92
  Satisfied | 73
  Unsatisfied | 3
  Very unsatisfied | 1

8. Secondary Outcome: Number of Participants for Physicians' Assessment of Efficacy
Description: Subjective assessment by the physician to evaluate control of bleeding. Physician rated assessment could be categorized as Very good, Good, Moderate, or Poor; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 269
participants
  Very good | 111
  Good | 111
  Moderate | 38
  Poor | 9

9. Secondary Outcome: Number of Participants for Patients' Assessment of Efficacy
Description: Subjective assessment by the participant to evaluate control of bleeding. Patient rated assessment could be categorized as Very good, Good, Moderate, Poor, or No specification; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 269
participants
  Very good | 103
  Good | 116
  Moderate | 35
  Poor | 11
  No specification | 4

10. Secondary Outcome: Number of Participants for Physicians' Assessment of Tolerance
Description: Subjective assessment by the physician to evaluate the participants' tolerance of treatment with ReFacto (i.e., dose, administration method, or adverse effects). Physician rated assessment could be categorized as Very good, Good, Moderate, or Poor; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 269
participants
  Very good | 130
  Good | 137
  Moderate | 2

11. Secondary Outcome: Number of Participants for Patients' Assessment of Tolerance
Description: Subjective assessment by the participant to evaluate tolerance of treatment with ReFacto (i.e., dose, administration method, or adverse effects). Patient rated assessment could be categorized as Very good, Good, Moderate, Poor, or No specification; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 269
participants
  Very good | 131
  Good | 132
  Moderate | 1
  Poor | 1
  No specification | 4

12. Secondary Outcome: Number of Participants for Physicians' Assessment of Handling of ReFacto
Description: Subjective assessment by the physician to evaluate the participants' handling (preparation and administration) of ReFacto. Physician rated assessment could be categorized as Very good, Good, Moderate, or Poor; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 269
participants
  Very good | 109
  Good | 154
  Moderate | 6

13. Secondary Outcome: Number of Participants for Patients' Assessment of Handling of ReFacto
Description: Subjective assessment by the participant on handling (preparation and administration) of ReFacto. Patient rated assessment could be categorized as Very good, Good, Moderate, Poor, or No specification; no criteria was pre-specified for the assessment categories in this observational study.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 269
participants
  Very good | 99
  Good | 154
  Moderate | 11
  Poor | 1
  No specification | 4

14. Secondary Outcome: Number of Participants for Days of Sick Leave Per Month
Description: Days of sick leave (missing work or school) per month categorized as No days of absence, Number of days of absence, Long-term inability to work or study, Not employed or at school, or No specification.
Time Frame: Baseline up to a mean duration of 54 months
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | ReFacto (Moroctocog Alfa)
Number analyzed (Participants) | 169
participants
  No days of absence | 87
  <6 days of absence | 32
  6 to 10 days of absence | 4
  >10 days of absence | 8
  Long-term inability to work or study | 0
  Not employed or at school | 36
  No specification | 2

ADVERSE EVENTS:
Time Frame: Baseline up to a mean duration of 54 months
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | ReFacto (Moroctocog Alfa)
Serious Adverse Events (participants affected / at risk) | 141/288
Other Adverse Events (participants affected / at risk) | 118/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReFacto (Moroctocog Alfa) (N=288)
Haemolysis (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 2
Conductive deafness (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal infarction (Gastrointestinal disorders) | 1
Lip haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Concomitant disease progression (General disorders) | 1
Condition aggravated (General disorders) | 6
Death (General disorders) | 1
Developmental delay (General disorders) | 1
Drug ineffective (General disorders) | 42
Impaired healing (General disorders) | 1
Local swelling (General disorders) | 1
Medical device complication (General disorders) | 1
Pyrexia (General disorders) | 1
Thrombosis in device (General disorders) | 1
Unevaluable event (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Gallbladder polyp (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 3
Acquired immunodeficiency syndrome (Infections and infestations) | 1
Anogenital warts (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cerebral toxoplasmosis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 2
Implant site infection (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 2
Skull fractured base (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Anti factor VIII antibody positive (Investigations) | 1
Anti factor VIII antibody test (Investigations) | 22
Antiphospholipid antibodies (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Biopsy testes (Investigations) | 1
Blood urine present (Investigations) | 1
Catheterisation cardiac (Investigations) | 1
Coagulation factor VIII level decreased (Investigations) | 1
Coagulation factor inhibitor assay (Investigations) | 1
Drug specific antibody present (Investigations) | 1
Free haemoglobin present (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Investigation (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 8
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 4
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 5
Convulsion (Nervous system disorders) | 1
Cubital tunnel syndrome (Nervous system disorders) | 1
Dyspraxia (Nervous system disorders) | 1
Febrile convulsion (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Antisocial behaviour (Psychiatric disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Enuresis (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal haemorrhage (Renal and urinary disorders) | 1
Testicular haemorrhage (Reproductive system and breast disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Adenotonsillectomy (Surgical and medical procedures) | 1
Arthrodesis (Surgical and medical procedures) | 1
Bone operation (Surgical and medical procedures) | 1
Central venous catheter removal (Surgical and medical procedures) | 4
Dental care (Surgical and medical procedures) | 1
Ear tube insertion (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Joint arthroplasty (Surgical and medical procedures) | 2
Joint surgery (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 2
Ossiculoplasty (Surgical and medical procedures) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 2
Thyroidectomy (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Vascular operation (Surgical and medical procedures) | 1
Wisdom teeth removal (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 1
Haematoma (Vascular disorders) | 7
Haemorrhage (Vascular disorders) | 9
Vein disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReFacto (Moroctocog Alfa) (N=288)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 3
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Cheilosis (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Lip haemorrhage (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Tooth loss (Gastrointestinal disorders) | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Discomfort (General disorders) | 1
Drug ineffective (General disorders) | 2
General physical health deterioration (General disorders) | 1
Inflammation (General disorders) | 2
Influenza like illness (General disorders) | 3
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 3
Pyrexia (General disorders) | 6
Unevaluable event (General disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 3
Acquired immunodeficiency syndrome (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
HIV infection (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media viral (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Accident at work (Injury, poisoning and procedural complications) | 1
Bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Electric shock (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 18
Foot fracture (Injury, poisoning and procedural complications) | 1
Genital injury (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 5
Injury (Injury, poisoning and procedural complications) | 5
Joint injury (Injury, poisoning and procedural complications) | 6
Joint sprain (Injury, poisoning and procedural complications) | 2
Limb crushing injury (Injury, poisoning and procedural complications) | 3
Limb injury (Injury, poisoning and procedural complications) | 8
Mouth injury (Injury, poisoning and procedural complications) | 2
Muscle rupture (Injury, poisoning and procedural complications) | 1
Open wound (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 5
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 4
Wound (Injury, poisoning and procedural complications) | 3
Arthroscopy (Investigations) | 1
Biopsy stomach (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Blood urine present (Investigations) | 1
Coagulation factor VIII level decreased (Investigations) | 10
Endoscopy upper gastrointestinal tract (Investigations) | 1
Free haemoglobin present (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 37
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Lordosis (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disturbance in attention (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Mental impairment (Nervous system disorders) | 1
Tongue biting (Nervous system disorders) | 2
Affect lability (Psychiatric disorders) | 1
Apathy (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Violence-related symptom (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Renal haemorrhage (Renal and urinary disorders) | 3
Renal pain (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Breast haematoma (Reproductive system and breast disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Adenotonsillectomy (Surgical and medical procedures) | 1
Bursa removal (Surgical and medical procedures) | 1
Catheterisation venous (Surgical and medical procedures) | 1
Central venous catheter removal (Surgical and medical procedures) | 2
Central venous catheterisation (Surgical and medical procedures) | 4
Dental care (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 3
Joint injection (Surgical and medical procedures) | 1
Medical device implantation (Surgical and medical procedures) | 1
Medical device removal (Surgical and medical procedures) | 1
Penile operation (Surgical and medical procedures) | 1
Plastic surgery (Surgical and medical procedures) | 1
Radiotherapy to joint (Surgical and medical procedures) | 2
Suture insertion (Surgical and medical procedures) | 1
Suture removal (Surgical and medical procedures) | 1
Synovectomy (Surgical and medical procedures) | 2
Tonsillectomy (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 5
Wisdom teeth removal (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 9
Haemorrhage (Vascular disorders) | 22
Lymphostasis (Vascular disorders) | 1
Unevaluable event (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.